CLINICAL TRIAL: NCT01657084
Title: Stopping and Preventing Epileptic Seizures Using a Partial Rebreathing Mask
Acronym: EpiCapno
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012051485
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tonic-clonic seizures (Experimental): Patients with tonic-clonis seizures are observed in a video/EEG room. In the case of seizures, the treatment mask or dummy mask are administered, according to a randomized cross-over study design.
  Interventions: Device: CDA Mask; Device: Dummy mask
- Generalized Paroxysms (Experimental): Patients with generalized epileptic paroxysms are observed by EEG during baseline, treatment mask and dummy mask use, according to a randomized cross-over study design.
  Interventions: Device: CDA Mask; Device: Dummy mask
- Group 3 (Experimental): Patients with epileptic paroxysms are observed by EEG during baseline, treatment mask and dummy mask use, according to a randomized cross-over study design.
  Interventions: Device: CDA Mask; Device: Dummy mask

INTERVENTIONS:
Device: CDA Mask — The CDA (Carbon Dioxide Accumulation) mask effectuates an increase in the inspired CO2 fraction, while allowing an adequate supply of fresh air to the patient.
Device: Dummy mask — The dummy mask is similar in appearance to the treatment mask, but causes only a negligible change in blood gases

SUMMARY:
By enabling a partial rebreathing of expired gas, a moderate respiratory acidosis is induced, without causing hypoxia in the patient.

Based on the scientific literature on the subject, the study hypothesis is that the fall in body pH will be able to stop and/or prevent epileptic brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy
* 18-80 years

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Length of epileptic seizure (subgroup 1) | Duration of mask treatment during acute seizures: approx. 3 minutes from start of mask treatment until end of seizure
  Length of epileptic seizure with treatment mask vs. dummy mask
Frequency of epileptic paroxysms (subgroups 2 and 3) | Duration of mask treatment: 45 minutes (group 2) or 10 minutes (group 3) during which patient is monitored with EEG
  Frequency of epileptic paroxysms as measured by EEG, treatment mask vs. dummy mask

SECONDARY OUTCOMES:
Oxygen saturation during mask treatment | Duration of mask treatment
  Measures oxygen saturation using a pulse oximeter during mask treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Christensen, M.D., Ph.d., Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - The Epilepsy Hospital Filadelfia, Dianalund